CLINICAL TRIAL: NCT01664845
Title: Effects of Metformin, Pegylated Interferon Alpha and Ribavirin for Chronic Hepatitis C With Insulin Resistance
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wei-Lun Tsai, Attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS12-CT3-16
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Hepatitis c; Insulin Resistance
Keywords: hepatitis c; metformin; pegylated interferon
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance; Hepatitis C | interventions — Metformin; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin, pegylated-IFN, ribavirin (Active Comparator): metformin,pegylated-IFN and ribavirin
  Interventions: Drug: metformin; Drug: pegylated-IFN; Drug: ribavirin
- Pegylated-IFN and ribavirin (Placebo Comparator): pegylated -IFN and ribavirin
  Interventions: Drug: pegylated-IFN; Drug: ribavirin

INTERVENTIONS:
Drug: metformin — metformin 500mg tid
  Other Names: glucophage
  Arms: metformin, pegylated-IFN, ribavirin
Drug: pegylated-IFN — pegasys 180 mcg qw
  Other Names: pegasys
Drug: ribavirin — ribavirin 800-1200 mg qd according to BW

SUMMARY:
The aim of the study is to investigate the treatment response of metformin, Peg-IFN and ribavirin combination therapy for chronic hepatitis C virus (HCV).

DETAILED DESCRIPTION:
Current standard of treatment for HCV with pegylated interferon(Peg-IFN)-alpha and ribavirin can achieve sustained virological response (SVR) in only 60-90% of patients. Insulin resistance is an important factor of non-response to combination therapy. Metformin is a insulin sensitizer and can effectively reduce insulin resistance. The aim of the study is to investigate the treatment response of metformin, Peg-IFN and ribavirin combination therapy for chronic HCV.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA (+) and ALT > 40 U/L
* Compensated liver
* HOMA-IR > 2

Exclusion Criteria:

* neutrophil <1500/mm3
* male: Hb < 13 g/dl, female: Hb < 12 g/dl
* platelet < 80,000 /mm3
* Cr > 2.5 mg/dl
* Alcohol use > 20 gm per day
* uncontrolled depression, thyroid disease, autoimmune disease
* Pregnancy
* Hepatocellular carcinoma
* allergy to interferon or ribavirin
* Diabetes
* HBV/HIV co-infection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
sustained virological response | 24 weeks after treatment is stopped
  HCV RNA negative 24 weeks after treatment is stopped

SECONDARY OUTCOMES:
change of HOMA-IR | Serial change of HOMA-IR at baseline, 4 weeks and 12 weeks after treatment
  Check Serial change HOMA-IR at baseline, 4 weeks and 12 weeks after treatment

OTHER OUTCOMES:
RVR | HCV RNA At 4 weeks
  HCV RNA At 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Lun Tsai, MD, Principal Investigator — Department of Gastroenterology, Kaohsoung Veterans General Hospital
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Taiwan